CLINICAL TRIAL: NCT01139632
Title: The Contribution of Lp-PLA2 Level to the Presence of Coronary Plaques in Patients With Non Alcoholic Fatty Liver Disease
Acronym: 0030-10
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Other Study IDs: 0030-10
Record Dates: First submitted 2010-06-06; First posted 2010-06-08 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2010-06

CONDITIONS: Nonalcoholic Fatty Liver Disease; Coronary Artery Disease
Keywords: NAFLD; lP-pla2; Coronary Arthery Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The most common cause of death in patients with NAFLD(Nonalcoholic Fatty Liver Disease) is CAD(Coronary Artery Disease). NAFLD patients have 65% more mortality than general population. The aim of the investigators study is to diagnose early coronary artery disease in NAFLD patient by measuring of PLA2. The investigators expect that PLA2 will higher in patients with patients with combination of CAD, unstable plaque and NAFLD.

DETAILED DESCRIPTION:
Background: The most common cause of death in patients with NAFLD(Nonalcoholic Fatty Liver Disease) is CAD(Coronary Artery Disease). NAFLD patients have 65% more mortality than general population. The aim of our study is to diagnose early coronary artery disease in NAFLD patient by measuring of PLA2.

Methods: 60 patients with chest pain and low to intermediate risk for coronary events will undergo Cardiac CT and blood test measurement of enzyme PLA2, markers of inflammation: CRP, MDA(Malondialdehide), Paraoxonase, FFA(Free Fatty Acids), TG(Triglycerids) will performed.

CAD is defined as a stenosis of more than 50% in at least one major coronary artery, unstable plaque defined as low attenuated plaque <30HU and fatty liver defined as difference in liver and spleen attenuation value -10HU by using CT.

Expected results : we expect that PLA2 will higher in patients with patients with combination of CAD, unstable plaque and NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at intermediate risk for significant CAD was admitted to the hospital with the diagnosis of chest pain or undergoing elective CT coronarography due to suspection of coronary artery disease.
2. Male and female 18years or older.
3. Able to provide written informed consent.

Intermediate Risk patients for having significant CAD is deﬁned as:

* chest pain or dyspnea in the presence of negative stress tests;
* the absence of chest pain but positive stress tests;
* the absence of chest pain and of positive stress tests but intermittent arrhythmias

Exclusion Criteria:

1. Acute coronary syndrome presentation:

   * ST segment deviation on ECG and/or
2. Cardiac troponin elevation.
3. Chest pain in combination with positive tests for myocardial ischemia
4. Hemodynamic instability on presentation.
5. Inability to write inform consent.
6. Age <18 years.
7. Participation in an investigational study within the previous 30days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients at intermediate risk for significant CAD was admitted to the hospital with the diagnosis of chest pain or undergoing elective CT coronarography due to suspection of coronary artery disease.
  2. Male and female 18years or older.
  Intermediate Risk patients for having significant CAD is deﬁned as:
  a - chest pain or dyspnea in the presence of negative stress tests; b - the absence of chest pain but positive stress tests; c - the absence of chest pain and of positive stress tests but intermittent arrhythmias.
  Age <18 years.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-01 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nimer Assy, MD, Principal Investigator — ZIV MEDICAL CENTER, SAFED ISRAEL
Locations (1):
- Ziv medical center liver unit, Safed, Israel, Israel